CLINICAL TRIAL: NCT07353450
Title: An Open-Label, Single Center Study Evaluating the Safety, Tolerability, and Immunogenicity of Cizutamig for Patients With Moderate to Severe Ulcerative Colitis
Brief Title: A Study of Cizutamig for Patients With Ulcerative Colitis
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CND106-RUJN-2
Record Dates: First submitted 2025-12-26; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Ulcerative Colitis (UC)
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A Study of Cizutamig for Patients with Ulcerative Colitis (Experimental): Cizutamig intravenous intervention
  Interventions: Biological: cizutamig

INTERVENTIONS:
Biological: cizutamig — Cizutamig will be dosed according to the protocol

SUMMARY:
A Study of Cizutamig for Patients with Ulcerative Colitis

DETAILED DESCRIPTION:
An Open-Label, Single Center Study Evaluating the Safety, Tolerability, and Immunogenicity of Cizutamig for Patients with Moderate to Severe Ulcerative Colitis

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years of age at the time of signing the informed consent form (ICF)
2. Have an established diagnosis of UC
3. Have current evidence of active moderate to severe UC.
4. Have current evidence of UC extending proximal to the rectum
5. Demonstrated intolerance or inadequate response to ≥ 1 biologic and/or other advanced therapies
6. Stable use of any of the following background therapy (alone or in combination) up to Day 1
7. Have documentation of:

   1. A surveillance colonoscopy (performed according to local standards) within 12 months of or during Screening, for patients with pancolitis of > 8 years duration, left-sided colitis of > 12 years duration, or primary sclerosing cholangitis; OR
   2. In patients for whom Inclusion Criteria 7a does not apply, up-to-date colorectal cancer surveillance (performed according to local standard), for patients with family history of colorectal cancer, personal history of increased colorectal cancer risk, age > 50 years, or other known risk factors -

Exclusion Criteria:1. Inadequate clinical laboratory parameters at Screening 2. Gastrointestinal disease 3. Patients with active infection 4. Receipt of or inability to discontinue any excluded therapies as specified in the protocol 5. Receipt of live vaccine within 4 weeks prior to Screening 6. History of progressive multifocal leukoencephalopathy 7. History of primary immunodeficiency or a hereditary deficiency of the complement system 8. Central nervous system (CNS) disease 9. Have presence of 1 or more significant concurrent medical conditions per investigator judgment 10. Have a diagnosis or history of malignant disease within 5 years prior to Screening 11. History of plasma cell dyscrasia 12. Need for uninterrupted anticoagulation 13. Serious mental illness, alcohol or drug abuse, dementia, or any other condition that would impair the patient's ability to receive the planned treatment or to understand informed consent at the study site as determined by local practice 14. Inability to comply with protocol-mandated requirements 15. History of severe allergic or anaphylactic reactions to mAb therapy or any constituents of cizutamig 16. History of severe allergic or anaphylactic reactions, or intolerance to required antimicrobial prophylaxis 17. History of or planned solid organ transplant and/or autologous or allogeneic hematopoietic stem cell transplantation for the duration of the study; or a corneal transplant within 12 weeks prior to Screening 18. Major surgery requiring use of general anesthesia within 12 weeks prior to Screening or planned or expected major surgery during the study period.

19. History of splenectomy, including patients with functional asplenia 20. Any serious medical condition or abnormality on clinical laboratory testing 21. Inability to comply with contraception requirements as specified in the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | Week 52
  1. Incidence of treatment-emergent adverse events (TEAEs) through end of study.
  2. Severity Grade of treatment-emergent adverse events (TEAEs) through end of study.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No